CLINICAL TRIAL: NCT01450319
Title: Phase II Clinical Study of Cetuximab in Refractory Colorectal Cancer With K-RAS Mutated and Favourable FcγR IIa (CD32) Genotype
Brief Title: Cetuximab in Refractory Colorectal Cancer With K-RAS Mutated and Favorable FcγRIIa (CD32) Genotype
Acronym: MUTEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck, S.L., Spain (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 062202-529; 2010-023580-18 (EudraCT Number)
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Neoplasms
Keywords: K-RAS; FcγRII/IIIa genotypes; CRC; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab (Experimental)
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Cetuximab will be administered intravenously at a dose of 500 milligram per square meter (mg/m^2) every 2 weeks until disease progression, death, or consent withdrawal.
  Other Names: Erbitux

SUMMARY:
This national, multicenter, open-label phase 2 study without any control arm aims to evaluate the activity of cetuximab monotherapy in the treatment of refractory colorectal cancer in subjects with K-RAS mutated and FcγRIIa polymorphism tumors, in which there is no therapeutic alternative for treatment. Failure of the first and second line conventional therapeutic lines was documented.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent form signed by the subject
* Age greater than or equal to (>=) 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (=<) 2
* Life expectancy of greater than (>) 2 months
* Histological confirmed colorectal cancer (CRC) with mutated K-RAS and favorable genotypes (any H in FcγRIIa-131). Selection will be done only based on Cluster of differentiation (CD)32 polymorphisms
* Epidermal growth factor receptor (EGFR) expression in his/her tumor sample
* Stage 4 metastatic disease, with at least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria, documented within 28 days prior to the study inclusion
* Tumor tissue sample available for the assessment of K-RAS status and FcγRIIa (CD32) genotype
* Subject who has received at least 2 prior therapeutic lines
* Adequate bone marrow function, defined as:

  * haemoglobin > 9.0 gram per deciliter (g/dL)
  * platelet count >100*10^9 per liter
  * absolute neutrophil count (ANC) >=1.5*10^9/Liter
* Adequate hepatic and renal function, defined as:

  * Serum bilirubin =<1.5 times the upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =<2.5*ULN in absence of liver metastasis and ALT and AST =<5*ULN in the presence of liver metastasis
  * Alkaline phosphatase =<2.5*ULN or =<5 in the presence of liver metastasis or =<10 in the absence of liver metastasis
  * Creatinine clearance >= 50 milliliter per minute (mL/min) (according to Cockcroft and Gault formula) or serum creatinine <1.5*ULN
* Adequate recovery after recent surgery, chemotherapy or radiotherapy. Prior major surgery, chemotherapy, treatment with an investigational product or radiotherapy must have occurred at least 4 weeks before study inclusion
* Women of child-bearing potential must have a negative pregnancy test performed within 7 days prior to the study inclusion. Postmenopausal women must be amenorrheic for at least 12 months. If the risk of conception exists both male and female subjects must use effective contraception (for example, abstinence, intrauterine device (IUD), oral contraceptive, double barrier method or to be surgically sterile) since the signature of the consent form until at least 6 months after the end of treatment or end of last dose, whichever occurs first

Exclusion Criteria:

* Previous treatment with monoclonal antibodies against EGFR
* Toxicity, due to previous treatment, not resolved to Grade 1 before the subject's inclusion into the study
* Clinically relevant coronary disease or myocardial infarction, unstable angina, Grade >=2 congestive cardiac insufficiency according to New York Heart Association (NYHA) within 6 months before starting the study treatment
* Clinically significant vascular disease (for example, aortic aneurysm which requires surgery, pulmonary embolism, recent peripheral arterial thrombosis) within 12 months prior to starting the study treatment
* Evidence of uncontrolled brain metastases
* History of active neurological disease
* History of uncontrolled seizures
* History of lung fibrosis, acute pulmonary damage or interstitial pneumonia
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C infection, or presence of severe, uncontrolled intercurrent infections or other severe uncontrolled concomitant diseases
* Current Grade >=2 (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE]) infection
* History of uncontrolled diabetes, uncontrolled hypertension or hepatic involvement
* Known or suspected allergy or hypersensitivity to cetuximab
* History of previous malignancy other than CRC occurring within 5 years before starting the study treatment, except for previously cured basal cell carcinoma of skin or carcinoma in situ of the cervix or urinary bladder treated more than 2 years before recruitment
* Participation in another treatment study with an investigational drug within the last 30 days
* Pregnancy or lactation
* Any medical, psychological, psychiatric or social uncontrolled problem which may interfere in the participation of the subject in the study or in the evaluation of the study results
* Psychological, familiar or geographic conditions not allowing the adequate follow-up and adherence to the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck, S.L., Spain
Locations (9):
- Spain (9):
  - Research Site, A Coruña
  - Research Site, Asturias
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Navarra
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Valencia

REFERENCES:
- [Derived] Manzanares-Martin B, Cebrian Aranda A, Del Puerto-Nevado L, Gonzalez R, Solanes S, Gomez-Espana MA, Garcia-Foncillas J, Aranda E. Improving selection of patients with metastatic colorectal cancer to benefit from cetuximab based on KIR genotypes. J Immunother Cancer. 2021 Apr;9(4):e001705. doi: 10.1136/jitc-2020-001705. PMID 33833048

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 73 subjects were enrolled in the trial. Out of 73 subjects, 70 subjects received the study drug and start the study and three subjects were excluded from the modified intent-to-treat (MITT) analysis set.
Groups:
- Cetuximab: Cetuximab was administered intravenously at a dose of 500 milligram per square meter (mg/m^2) every 2 weeks until disease progression, death, or consent withdrawal.
Period: Overall Study
Arm/Group | Cetuximab
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: MITT analysis set included all the subjects who received study drug treatment.
Arm/Group | Cetuximab
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.61 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Time
Description: Overall survival was defined as the time from date of informed consent signature until death.
Time Frame: From the date of informed consent signature until death, assessed up to 3 years
Population: MITT analysis set included all the subjects who received study drug treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cetuximab
Number analyzed (Participants) | 70
Months | 6.71 [5.42 to 8.05]

2. Secondary Outcome: Percentage of Subjects With Disease Control Rate (DCR)
Description: DCR was defined as those subjects achieving complete response (CR), partial response (PR) or stable disease (SD), according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v.1.1). For target lesions (TLs), CR was defined as the disappearance of all TLs; PR was defined as at least a 30 percent (%) decrease in the sum of longest diameter (SLD) of the TLs, taking as a reference the baseline (BL) SLD; Stable disease (SD) was defined as neither sufficient decrease in SLD to qualify for PR nor sufficient increase in SLD to qualify for PD; and PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since the treatment started. For non-target lesions (NTLs), CR was defined as the disappearance of all NTLs and normalization of tumor marker levels; SD was defined as the persistence of 1 or more NTLs and/or maintenance of tumor marker levels above normal limits; and progressive disease (PD) was defined as the appearance
Time Frame: From the date of informed consent signature until progressive disease, assessed up to 3 years
Population: MITT analysis set included all the subjects who received study drug treatment.
Measure: Number; unit: Percentage of subjects
Arm/Group | Cetuximab
Number analyzed (Participants) | 70
Percentage of subjects | 22.86

3. Secondary Outcome: Progression Free Survival (PFS) Time
Description: PFS was defined as the time from informed consent signature until PD or death, whatever occurred first. Subjects who did not have disease progression or were lost to follow-up, were censored at the date of last contact, known to be alive and progression free; moreover, those subjects who started a new treatment (different from cetuximab), were censored at the date of starting the new treatment. For TLs, PD was defined at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from BL or the appearance of one or more new lesions. For NTLs, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing NTLs. Participants without second-line PD or death were censored at the date of last tumor assessment where non-progression was documented.
Time Frame: From the date of informed consent signature until progressive disease (PD) or death, assessed up to 3 years
Population: MITT analysis set included all the subjects who received study drug treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cetuximab
Number analyzed (Participants) | 70
Months | 2.53 [2.43 to 2.70]

4. Secondary Outcome: Number of Subjects With Adverse Events (AEs), Serious Adverse Events (SAEs), AEs Leading to Discontinuation, AEs Leading to Death
Description: An AE was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A SAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the date of enrollment up to 30 days after the last dose of study drug administration, assessed up to 3 years
Population: Safety analysis set included all the subjects who received at least one dose of the study drug treatment.
Measure: Number; unit: Subjects
Arm/Group | Cetuximab
Number analyzed (Participants) | 70
Subjects
  AEs | 69
  SAEs | 17
  AEs leading to discontinuation | 2
  AEs leading to death | 3

5. Secondary Outcome: Number of Subjects With Fcγ Receptors (FCγR) IIa/IIIa Polymorphisms
Description: The antibody fragment C portion (FCy) of cetuximab interacts with Fc-gamma receptors (FCyRs) expressed by immune effector cells. Polymorphisms were described in genes coding for FCyRIIa and in FCyRIIIa. A histidine/arginine polymorphism at position 131 for FCyRIIa gene and valine ⁄ phenylalanine polymorphism at position 158 for the FCyRIIIa gene were reported to be functionally relevant in the ADCC mechanism. All subjects were analyzed and classified as carriers of every different polymorphism of FCy Receptors: for FCyRIIa (H/H, homozygous alleles with histidine and R/H, heterozygous alleles with arginine/histidine) and FCyRIIIa (V/V, homozygous alleles with valine, F/F, homozygous alleles with phenylalanine and F/V, heterozygous alleles with valine ⁄ phenylalanine) (units: subjects with every type of polymorphism) .The FCyR genotype was determined using a TaqMan Allelic Discrimination Assay.
Time Frame: Baseline
Population: MITT analysis set included all the subjects who received study drug treatment. Subjects may fall into more than one category.
Measure: Number; unit: Subjects
Arm/Group | Cetuximab
Number analyzed (Participants) | 70
Subjects
  FcγRIIa: H/H | 27
  FcγRIIa: R/H | 43
  FcγRIIIa: V/V | 6
  FcγRIIIa: F/F | 28
  FcγRIIIa: F/V | 36

6. Secondary Outcome: Overall Survival (OS) Related to Codon G13D
Description: OS was defined as the time from informed consent signature until death. Subjects without death were censored at the last date known alive (within the study).
Time Frame: From the date of informed consent signature until death, lost-to-follow-up or end of study, whatever occurred first (maximal up to 3 years)
Population: MITT analysis set included all the subjects who received study drug treatment. Here "Number of subjects analyzed" signifies total number of evaluable subjects for this outcome measure; "n" signifies number of evaluable subjects for each category, as specified.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab
Number analyzed (Participants) | 62
months
  G13D (n=14) | 7.2 [4.8 to NA] — Data could not be evaluated due to lack of events.
  No G13D (n=48) | 6.3 [4.8 to 7.9]

7. Secondary Outcome: Overall Survival (OS) Related to Killer Inhibitory Receptors 2DS4 (KIR2DS4) Functional Receptor (f/d) and Non-functional Receptor (NFR)
Description: as for outcome 6
Time Frame: From the date of informed consent signature until death, lost-to-follow-up or end of study, whatever occurred first (maximal assessed up to 3 years)
Population: MITT analysis set included all the subjects who received study drug treatment. Here "Number of subjects analyzed" signifies number of evaluable subjects for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab
Number analyzed (Participants) | 66
months
  f/d (n=10) | 4.8 [2.2 to 7.3]
  NFR (n=56) | 7.4 [6.0 to 8.4]

8. Secondary Outcome: Beta 2-microglobulin
Time Frame: Baseline, Week 8
Population: MITT analysis set included all the subjects who received study drug treatment. Here "n" signifies number of evaluable subjects for each category, as specified.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Cetuximab
Number analyzed (Participants) | 70
microgram per milliliter (mcg/mL)
  Baseline (n=61) | 2.35 (0.58)
  Week 8 (n=29) | 2.37 (1.13)

ADVERSE EVENTS:
Time Frame: AEs with onset from the date of enrollment up to 30 days after the last dose of study drug administration; assessed up to 3 years
Arm/Group | Cetuximab
Serious Adverse Events (participants affected / at risk) | 17/70
Other Adverse Events (participants affected / at risk) | 69/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=70)
Cholestaticjaundice (Hepatobiliary disorders) | 1
Acute cholecystitis (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Liver failure (Hepatobiliary disorders) | 1
Pyrexia (General disorders) | 1
Pain (General disorders) | 1
General malaise (General disorders) | 1
Catheter point infection (Infections and infestations) | 1
Listeria meningitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Heart failure (Cardiac disorders) | 1
Bowel obstruction (Gastrointestinal disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Acute renal failure (Renal and urinary disorders) | 1
Spontaneous hematoma (Blood and lymphatic system disorders) | 1
Pathologic fracture (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=70)
Rash (Skin and subcutaneous tissue disorders) | 39
Skin toxicity (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 8
Skin fissures (Skin and subcutaneous tissue disorders) | 8
Dermatitis (Skin and subcutaneous tissue disorders) | 8
Acne (Skin and subcutaneous tissue disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 6
Asthenia (General disorders) | 32
Mucosal inflammation (General disorders) | 10
Pyrexia (General disorders) | 10
Oedema peripheral (General disorders) | 6
Pain (General disorders) | 5
Constipation (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 9
Abdominal pain upper (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 16
Hypomagnesaemia (Metabolism and nutrition disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Catarrh (Respiratory, thoracic and mediastinal disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 9
Insomnia (Psychiatric disorders) | 5
Jaundice (Hepatobiliary disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other